CLINICAL TRIAL: NCT05356663
Title: Comparative Effects of Hold Relax Technique and Mulligan Mobilization on Pain, ROM and Function in Post Operative Knee Joint: A Randomised Controlled Trail
Brief Title: Comparative Effects of Hold Relax Technique and Mulligan Mobilization in Post Operative Knee Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0110 Imbesat
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Pain
Keywords: mulligan mobilization with movement; post-operative knee joint; hold relax technique; knee stiffness; range of motion
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization with movement (Experimental): Mulligan Mobilization with movement + Baseline treatment (Moist Heat Pack) Group will receive mulligan mobilization with movement with the frequency of 3 sets and 10 repetitions 3 times a week for 6 weeks.
  Interventions: Other: Mulligan Mobilization
- Hold relax technique (Experimental): Hold relax technique + Baseline treatment (Moist Heat Pack) Group will receive Hold Relax Technique of PNF included, 5 repetitions will be given 3 times/week for 6 weeks.
  Interventions: Other: Hold Relax

INTERVENTIONS:
Other: Mulligan Mobilization — Medial glide MWM for knee flexion (supine) Lateral glide MWM for knee flexion (supine) Medial glide MWM for knee flexion.( prone ) Lateral glide MWM for knee flexion (prone)
  Arms: Mulligan Mobilization with movement
Other: Hold Relax — Hold-relax technique of PNF included, the affected knee will be flexed passively to the end of range with the therapist's hand on the patient's lower leg. Patients then performed 5 s of quadriceps contraction against the resistance of the therapist. Patients will be asked not to let move. At the end of 5 s, the patients will be asked to totally relax for 10 s and the therapist pushed the knee into more flexion and hold at that newly acquired range
  Arms: Hold relax technique

SUMMARY:
The aim of this study is to investigate the comparative effects of hold relax technique and mulligan mobilization on pain, ROM and function in post operative knee joint.

DETAILED DESCRIPTION:
Stiffness or restricted ROM of the knee joint is a term used commonly to describe any traumatic condition occurring within or around the knee joint. It can result from direct and indirect below and is experienced as pain with activity, local tenderness to palpation, and decreased ability to tolerate tension, which results in decreased movement and functional strength. Post-traumatic knee stiffness and loss of range of motion is a common complication of injuries to the knee area. Immobilization of human knees for several weeks or more can result in stiffness and loss of range of motion in the joints. After knee arthroplasties, cruciate ligament repairs and trauma may lead to contracture of muscles and knee instability. Limitations of joint movements both flexion and extension suggests intraarticular pathology.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female of age 20 to 40 years

  * Knee pain 3 or more on VAS
  * Patients with grade 3 or more than 3 power of knee muscle
  * Subjects with post traumatic stiffness of knee joint having a minimum of 70 degree of knee flexion

Exclusion Criteria:

* Hypermobile and unstable joint

  * Soft tissue injuries
  * Joint infection and loosening
  * Other complication of post fracture/ TK

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | 3 months
  The most common validated tool for assessment of pain in clinical tests is the numeric pain rating score (NPRS), a 10-point scale where 0 indicates no pain and 10 indicates severe pain
Goniometer for Range of motion | 3 months
  It is a technique in which instrument named as goniometer purports to measure accurately the movements present in a simple or composite joint. Actually a goniometer is not used so much to measure the exact number of degrees of the movement in the joint as to find out whether there is increase or decrease of such movements. In order to do this, it is desirable that a goniometer should provide an easy method of reference to the joint or joint being examined and also provide a fixed base line point from which to measure any increase or decrease of movement
Time up and go test for functional ability | 3 months
  The test consists of measuring the time it takes for an individual to get up from the chair and walk as fast as possible to a 3-meter walk, turn around, come back and sit down. Time taken to complete the test were measured on stopwatch to the nearest 1/100 of the second

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Govt. Hospital DHQ, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No